CLINICAL TRIAL: NCT03237585
Title: Impact Assessment of the Rural Response System to Reduce Violence Against Women in Ghana
Acronym: GhanaCHiPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: University of Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC031-9/2015
Record Dates: First submitted 2017-07-01; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Domestic Violence; Physical Violence; Sexual Violence
Keywords: gender based violence; violence against women; intimate partner violence; impact assessment; rural response system; cluster randomised controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i) Intervention arm- Receive Gender Centre's RRS package (Experimental)
  Interventions: Behavioral: Rural response system (RRS) intervention to reduce violence against women
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Rural response system (RRS) intervention to reduce violence against women — The Rural Response System which uses the strategy of trained community members known as Community-based action team, COMBAT to undertake awareness-raising on gender-based violence as well as providing support to victims of violence to access justice and other relevant services.
  Arms: i) Intervention arm- Receive Gender Centre's RRS package

SUMMARY:
AIM: To assess the community level impact of the Gender Centre's Rural Response System (RRS) in reducing violence against women (VAW) in Ghana.

METHODS:

Design: An unmatched cluster randomised controlled trial with two arms i) Intervention arm- Receive Gender Centre's RRS /COMBAT package for communities as well as state agencies. Control arm - No intervention. Qualitative component Setting: Rural and urban communities in the Central Region of Ghana. i). Rural and urban communities in four (4) Districts located in the Central Region of Ghana. Two districts are along the Coast (Abura and Komenda) while the other two (Agona and Upper Denkyira) are inland districts.

ii). State Agencies (DOVVSU/Police, CHRAJ, Social Welfare, and Health Services).

Interventions: Carried out in two Districts - Agona district and Komenda district. Workings of the intervention arm will be facilitated by the Gender Studies and Human Rights Documentation Centre in Ghana.

Sample size: A total of 3280 adults (1640 women and 1640 men) from 20 clusters per trial arm (approximately 82 households per cluster) will be recruited at baseline and again at post-intervention survey. Sampling format will be a community survey with independent samples design (i.e. in each community, the people surveyed at baseline may not necessarily be the same people who are surveyed at post intervention. Clusters refer to the selected localities and their participating communities in each district.

Evaluation design: Pre-test all study participants with a standardized instrument then introduce the independent variable (intervention) to the experimental group while withholding it from the control group. After 24 months of intervention, post-test both groups with the same instrument and under the same conditions as the pretest (baseline). Compare the amount of change in dependent variable for both experimental and control groups.

Data analysis: The data will be analysed by intention to treat. The past 12 months prevalence of IPV will be compared between arms in the study.

DETAILED DESCRIPTION:
The Rural Response System (RRS) was a strategy developed by the Gender Centre over a decade ago to deal with the major problems related to VAW including poor institutional response to VAW; high degree of tolerance of VAW in the Ghanaian society which is perpetuated by strong perceptions that domestic violence is a private matter; the general confusion about what constitutes violence and ignorance about the causes, consequences and mechanisms that perpetuate VAW [1]. It is generally acknowledged that to enable victims to take advantage of laws and policies for their protection, there is the need to have structures in place that support and enable them assert their rights. The RRS model uses multiple strategies (such as training, sensitization and awareness-raising, support services, networking and coalition building, advocacy) targeting multiple stakeholders including women, men, religious and traditional leaders, policy makers, state agencies etc. to ensure that women are empowered to become their own agents of change, with communities that support and uphold women's rights and a state where gender sensitive laws and policies are implemented.

The Rural Response System uses the strategy of trained community members known as Community-based action team, COMBAT to undertake awareness-raising on gender-based violence as well as providing support to victims of violence to access justice. The RRS is stressed as a community initiative facilitated by GC to ensure community ownership. The selection of the COMBAT, the criteria for their selection and their roles are done by the community members with the GC serving only as a facilitator in this process. Teams usually work as a group when undertaking community sensitization and awareness-raising but could also work individually as they are encouraged to use every opportunity, such as community festivals and meetings, membership meetings of social associations, religious groupings, meetings of family and friends to carry out this role. The sensitization will be an ongoing process and not a one-off activity.

Goal and Objectives: Our project goal is to reduce the prevalence of VAW and promote and protect the rights of women and girls. We will do this by increasing the visibility of VAW as a social issue, improving the public's knowledge and understanding of the negative impact of VAW on the status of women and girls; establish a community based response system for the support and protection of women and provide counselling services as well as work with state agencies to ensure effective response to victims; whilst sharing best practice and key lessons learnt with other stakeholders.

With regard to the RRS model/COMBAT, the specific objectives of the impact assessment will be as follows: To assess the impact of the RRS model/COMBAT in reducing VAW; To determine whether RRS model/COMBAT interventions are effective in enabling women in to reduce their exposure to intimate partner violence (IPV) and men to reduce their perpetration of IPV; To assess if the RRS model changes discriminatory social norms and gender roles which consider VAW acceptable; To assess the extent to which RRS has changed individual attitudes about gender inequality To assess state institutional response to reported cases of VAW ;To assess whether the RRS model facilitated a shift in power relations between men and women in the household/community to become more equitable.

Study Setting: This study will be carried out in 4 Districts located in the Central Region of Ghana. Two districts are along the Coast (Abura and Komenda) while the other two (Agona and Upper Denkyira) are inland districts.

Study Population: Participating districts from the Central Region of Ghana were selected on the basis of operational and program considerations. Selection of districts was done using a census map of the Central Region that showed Inland and Coastal districts [2]. After excluding some districts on the grounds that previous intervention work on GBV has been carried out in those districts, two inland and two coastal districts were then purposively selected as study sites. Designated sites are separated from each other by a geographical buffer (at least one district wide) to reduce the possibility of intervention diffusing into control districts.

Sample Size Estimation: Sample size for a cluster randomized control trial in a community was defined at two levels: The level of randomization - number of clusters randomized, and the level of data collection - number of individuals surveyed in each household. Using the method of Hayes and Bennet [3], we estimated sample size (i.e. the number of clusters required in each arm of treatment) for an unmatched cluster-randomized control trial. The calculation made the following assumptions: Power: 90%; Ho (Pi_0): Proportion in the population that experience any form of IPV (emotional, physical, sexual violence, or all three forms). This estimate is based on national level data from the 2008 Ghana Demographic and Health Survey which indicates that among ever-married women age 15-49 years, 34.9% have experienced violence (any form) commuted by their husband/partner in the 12 months preceding the DHS survey [4]. Alpha (ɑ) = 0.05 (two-sided). K: coefficient of variation = 20%. This refers to the coefficient of variation between clusters for the outcome measure. We used k = 0.20 on the basis of district level census within the Central Region of Ghana [2]. We will oversample by 15% to allow for incomplete questionnaires. A total sample size of 1640 women and 1640 men will to be sampled from 20 clusters per trial arm. This would imply 90% power to detect a significant change at the 5% level with a 20% reduction in IPV incidence.

To randomize the districts, the names of the two Inland districts were written on a piece of paper and put in a bag. One paper was blindly drawn from the bag, the selected district was assigned as an intervention district, and the other designated as the control district. Clusters in the Ghana DHS are census listed localities with each locality comprising one or more enumeration areas. Owing to the nature of intervention design, participants will not be blind to their study arm. All clusters will be allocated numbers and the randomization done using a system of numbers. Within each selected district, lists of localities will be obtained from the Ghana Statistical Service, and a random sample of 10 localities from each district taken using simple random sampling.

Qualitative Approach: The qualitative approach will be adopted to provide in-depth understanding of the effects of the CHiPs intervention, if any, at individual, community as well as institutional levels. Qualitative methods will be used to assess the overall goal of the project; specifically evaluating the level of visibility for violence against women (VAW) issues in communities, knowledge and awareness of VAW and its outcomes. In this regard, various qualitative data collection techniques (Focus Group Discussions (9), In-depth Interviews (60), Key Informant Interviews (8) and Document Reviews will be used at baseline, midpoint (9 months) and the endpoint of the intervention (18 months) to collect data in both intervention and control communities. These will involve community members, COMBAT members, as well as critical stakeholders to examine community experiences, programmatic perspectives and outcomes as well as institutional responses.

At the individual level the Community FGDs and IDIs will explore knowledge about VAW, experiences with the intervention including Gender attitudes, Women's subordination, Tolerance of VAW, Social stigma for the victims of VAW, Decision making on number of children and spacing and Decision making on the use of contraceptives. FGDs with COMBAT Members will also explore themes on attitudes of service providers, Increased knowledge of community members on the impact of VAW, Perceptions about intervention and Assessment of the effectiveness of the programme. KIIs will assess Institutional response to VAW, Relevant laws on VAW, Women & societal responses to VAW, Improved institutional response to cases of VAW reported to State Agencies, and Institutional assessment of VAW cases.

Ethical Considerations: This research proposal is structured in accordance with the ethical principles provided by the World Medical Association Declaration of Helsinki (last updated in 2013) [5], and the Belmont report (1979) [6]. These documents emphasize respect for person's autonomy, justice, beneficence, and non-maleficence (do no harm) in the conduct of research with human participants. Ethical approval for the study will be sought from the Institutional Review Board at the Noguchi Memorial Institute for Medical Research, University of Ghana, and the South African Medical Research Council's Ethics Committee. This trial has been designed to ensure that the project does not expose participants to more than minimal risk (more than everyday risk). The study design has measures in place to minimize the potential of harm to participants and be able to respond to any adverse consequences i.e. emotional or psychological harm that may result from the questions that will be asked in this study. The following measures will be put in place to ensure that the study is conducted in an ethical correct manner. Complete privacy is essential for ensuring the security of the respondent and the interviewer. Asking about or reporting violence, especially in households where the perpetrator may be present at the time of interview, carries the risk of further violence. Accordingly, interviewers will be provided specific training for implementing the domestic violence module to enable the field staff to collect violence data in a secure, confidential, and ethical manner.

Informed Consent and Confidentiality: All research participants will be asked to give written informed consent before participating. Prospective participants will be informed of the purpose of the trial, procedures involved, risk and benefits of the trial and their rights as participants. All prospective participants will be informed that participation in the trial is voluntary, and that they may withdraw at any stage, or skip any question in the research with no adverse consequences to them. All participants will be assured that the information they provide in the trial will be handled confidentially and that findings will be reported with complete anonymity. Participants will be guaranteed that all the information collected will be kept confidential. The confidentiality of information given by participants will be ensured using codes on the questionnaires instead of subject names.

The study will be conducted over 36 months with recruitment commencing soon after ethical approvals have been granted. There will be one baseline survey, followed by 18 months of intervention, and one impact evaluation survey. This research is funded by the United Kingdom Government's Department for International development (DFID).

ELIGIBILITY:
Inclusion Criteria:

* Adult women (ages 18 to 49 years) and adult men (≥ 18 years) in the Central Region of Ghana
* Usually live (sleep and eat) in the household, have lived in the community for at least a year

Exclusion Criteria:

* Minor
* Not able to provide informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3280 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Past year incidence of intimate partner violence | 1 year
  The primary outcome indicator for this impact assessment is past year incidence of IPV (perpetration of physical and/or sexual IPV for men and experience for women).

SECONDARY OUTCOMES:
Institutional assessment of violence against women cases | 3 years
  Assess reported cases of violence against women

CONTACTS AND LOCATIONS:
Overall Officials: Richard Adanu, PhD, Principal Investigator — University of Ghana
Locations (1):
- Rural and Urban Communities, Abura, Komenda, Agona, Upper Denkyira, Central Region, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be published.
Supporting Information: Study Protocol
Time Frame: 2017
Access Criteria: Published in Open Access Journal

REFERENCES:
- [Background] 1. Gender Studies and Human Rights Documentation Centre, Breaking the Silence and Challenging the Mythos of Violence against Women and Children in Ghana. Report of a national study on Violence. Edited by Dorcas Coker-Appiah and Kathy Cusack. Gender and Human Rights Documentation Centre, 1998.
- [Background] 2. Ghana Statistical Service (GSS). 2013. 2010. Population and Housing Census, Regional Analytical Report; Central Region, Ghana: Ghana Statistical Service, Accra.
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] 4. Ghana Statistical Service (GSS), Ghana Health Service (GHS), and ICF Macro. 2009. Ghana Demographic and Health Survey 2008. Accra, Ghana: GSS, GHS, and ICF Macro.
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Department of Health, Education, and Welfare; National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research. The Belmont Report. Ethical principles and guidelines for the protection of human subjects of research. J Am Coll Dent. 2014 Summer;81(3):4-13. PMID 25951677